CLINICAL TRIAL: NCT02822326
Title: CD19-CAR-T2 Cells for Relapse/Refractory CD19 Positive Acute Leukemia-a Phase I Trial
Brief Title: Phase I Study of CD19-CAR-T2 Cells for Patients With Chemotherapy Resistant or Refractory CD19+ Acute Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government); Guangdong Zhaotai InVivo Biomedicine Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.GDREC2016198H
Record Dates: First submitted 2016-06-28; First posted 2016-07-04 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Acute Leukemia
Keywords: Leukemia; CART CD19; Chemotherapy Resistant; Chemotherapy Refractory; CD19 +; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD19-CAR-T2 T Cells (Experimental): The subject's T cells will be modified to those which could identify and kill the tumor cells (CD19+ cells). These CD19-CAR-T2 T cells will be infused over 10-15 minutes on days Day 1, 2 and 3 tentatively according to the response to infusion.
  Interventions: Biological: CD19-CAR-T2 Cells

INTERVENTIONS:
Biological: CD19-CAR-T2 Cells

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of chimeric antigen receptor 19 (CD19-CAR-T2 Cells) infusions in patients with chemotherapy resistant or refractory CD19+ acute Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed and/or refractory CD19 positive B-cell acute leukemia
* Eastern Cooperative Oncology Group (ECOG) performance status 《 3
* ALT/ AST 《 3x normal
* Bilirubin < 2.0 mg/dl
* Creatinine < 2.5 mg/dl and less than 2.5x normal for age
* LVEF》 45%
* Accept white blood cell collection
* Provide informed consent

Exclusion Criteria:

* Previous treatment with investigational gene or cell therapy medicine products
* Solitary extramedullary relapse
* Active hepatitis B , hepatitis C or HIV infection
* Uncontrolled active infection
* Presence of grade 2-4 acute or extensive chronic GVHD
* Active CNS involvement: epilepsy, paresis, aphasia, stroke, severe head trauma,
* Dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, uncontrolled mental illness, etc.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Received non-diagnostic purposes major surgery within the past 4 weeks
* Participated in any other clinical study within the past 4 weeks
* Used murine biological products (except blinatumomab), unless it is proved no anti-mouse antibodies exist.
* Pregnancy or breast-feeding women
* Use of prohibited drugs:
* Steroids: Therapeutic doses of steroids must be stopped > 72 hours prior to CD19-CAR-T2 Cells infusion
* Allogeneic cellular therapy: Any donor lymphocyte infusions (DLI) must be completed > 4 weeks prior to CD19-CAR-T2 Cells infusion
* GVHD therapies: Any drug used for GVHD must be stopped > 4 weeks prior to CD19-CAR-T2 Cells infusion
* Chemotherapy: i. The following drugs must be stopped > 1 week prior to CTL019 infusion and should not be administered concomitantly or following lymphodepleting chemotherapy: hydroxyurea, vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate <25 mg/m2, cytosine arabinoside < 10 mg/m2/day, asparaginase; ii. The following drugs must be stopped > 4 weeks prior to CTL019 infusion: salvage chemotherapy (e.g. clofarabine, cytosine arabinoside > 100 mg/m2, anthracyclines, cyclophosphamide), excluding the required lymphodepleting chemotherapy drugs
* Any situation that may increase the risk of the test or interfere with the test results

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose(MTD) of CD19 positive relapsed/ refractory acute leukimia treated wtih CD19-CAR-T2 cells | 24 weeks

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 12 months
  Adverse events and laboratory abnormalities (type, frequency and severity)
Overall Response Rate | 12 months
  Overall Response Rate (ORR), which includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi), as determined by assessments of peripheral blood, bone marrow, CNS symptoms, physical exam (PE) and CSF. The primary endpoint will be based on the IRC assessment. The local investigator's assessed results will be used for sensitivity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyu Weng, Dr., Principal Investigator — Guangdong Provincial People's Hospital; Peilong Lai, Dr., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunger SP, Lu X, Devidas M, Camitta BM, Gaynon PS, Winick NJ, Reaman GH, Carroll WL. Improved survival for children and adolescents with acute lymphoblastic leukemia between 1990 and 2005: a report from the children's oncology group. J Clin Oncol. 2012 May 10;30(14):1663-9. doi: 10.1200/JCO.2011.37.8018. Epub 2012 Mar 12. PMID 22412151
- [Background] Raetz EA, Bhatla T. Where do we stand in the treatment of relapsed acute lymphoblastic leukemia? Hematology Am Soc Hematol Educ Program. 2012;2012:129-36. doi: 10.1182/asheducation-2012.1.129. PMID 23233571
- [Background] Pulte D, Redaniel MT, Jansen L, Brenner H, Jeffreys M. Recent trends in survival of adult patients with acute leukemia: overall improvements, but persistent and partly increasing disparity in survival of patients from minority groups. Haematologica. 2013 Feb;98(2):222-9. doi: 10.3324/haematol.2012.063602. Epub 2012 Aug 28. PMID 22929974
- [Background] Schrappe M, Hunger SP, Pui CH, Saha V, Gaynon PS, Baruchel A, Conter V, Otten J, Ohara A, Versluys AB, Escherich G, Heyman M, Silverman LB, Horibe K, Mann G, Camitta BM, Harbott J, Riehm H, Richards S, Devidas M, Zimmermann M. Outcomes after induction failure in childhood acute lymphoblastic leukemia. N Engl J Med. 2012 Apr 12;366(15):1371-81. doi: 10.1056/NEJMoa1110169. PMID 22494120
- [Background] Forman SJ, Rowe JM. The myth of the second remission of acute leukemia in the adult. Blood. 2013 Feb 14;121(7):1077-82. doi: 10.1182/blood-2012-08-234492. Epub 2012 Dec 14. PMID 23243288
- [Background] Jensen MC, Popplewell L, Cooper LJ, DiGiusto D, Kalos M, Ostberg JR, Forman SJ. Antitransgene rejection responses contribute to attenuated persistence of adoptively transferred CD20/CD19-specific chimeric antigen receptor redirected T cells in humans. Biol Blood Marrow Transplant. 2010 Sep;16(9):1245-56. doi: 10.1016/j.bbmt.2010.03.014. Epub 2010 Mar 19. PMID 20304086
- [Background] Savoldo B, Ramos CA, Liu E, Mims MP, Keating MJ, Carrum G, Kamble RT, Bollard CM, Gee AP, Mei Z, Liu H, Grilley B, Rooney CM, Heslop HE, Brenner MK, Dotti G. CD28 costimulation improves expansion and persistence of chimeric antigen receptor-modified T cells in lymphoma patients. J Clin Invest. 2011 May;121(5):1822-6. doi: 10.1172/JCI46110. Epub 2011 Apr 11. PMID 21540550
- [Background] Chimeric Antigen Receptor-Modified T Cells in Chronic Lymphoid Leukemia; Chimeric Antigen Receptor-Modified T Cells for Acute Lymphoid Leukemia; Chimeric Antigen Receptor T Cells for Sustained Remissions in Leukemia. N Engl J Med. 2016 Mar 10;374(10):998. doi: 10.1056/NEJMx160005. No abstract available. PMID 26962747
- [Background] Porter DL, Hwang WT, Frey NV, Lacey SF, Shaw PA, Loren AW, Bagg A, Marcucci KT, Shen A, Gonzalez V, Ambrose D, Grupp SA, Chew A, Zheng Z, Milone MC, Levine BL, Melenhorst JJ, June CH. Chimeric antigen receptor T cells persist and induce sustained remissions in relapsed refractory chronic lymphocytic leukemia. Sci Transl Med. 2015 Sep 2;7(303):303ra139. doi: 10.1126/scitranslmed.aac5415. PMID 26333935
- [Background] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870
- [Background] Kochenderfer JN, Dudley ME, Kassim SH, Somerville RP, Carpenter RO, Stetler-Stevenson M, Yang JC, Phan GQ, Hughes MS, Sherry RM, Raffeld M, Feldman S, Lu L, Li YF, Ngo LT, Goy A, Feldman T, Spaner DE, Wang ML, Chen CC, Kranick SM, Nath A, Nathan DA, Morton KE, Toomey MA, Rosenberg SA. Chemotherapy-refractory diffuse large B-cell lymphoma and indolent B-cell malignancies can be effectively treated with autologous T cells expressing an anti-CD19 chimeric antigen receptor. J Clin Oncol. 2015 Feb 20;33(6):540-9. doi: 10.1200/JCO.2014.56.2025. Epub 2014 Aug 25. PMID 25154820
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Derived] Weng J, Lai P, Qin L, Lai Y, Jiang Z, Luo C, Huang X, Wu S, Shao D, Deng C, Huang L, Lu Z, Zhou M, Zeng L, Chen D, Wang Y, Chen X, Geng S, Robert W, Tang Z, He C, Li P, Du X. A novel generation 1928zT2 CAR T cells induce remission in extramedullary relapse of acute lymphoblastic leukemia. J Hematol Oncol. 2018 Feb 20;11(1):25. doi: 10.1186/s13045-018-0572-x. PMID 29458388